CLINICAL TRIAL: NCT04409522
Title: Evaluation of Therapeutic Effects of Melatonin by Inhibition of NLRP3 Inflammasome in COVID19 Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mohammad Sadegh Bagheri Baghdasht (Other)
Responsible Party: Sponsor-Investigator, Mohammad Sadegh Bagheri Baghdasht, Principal Investigator, Baqiyatallah Medical Sciences University
Organization: Baqiyatallah Medical Sciences University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IR.BMSU.REC.1399.039
Record Dates: First submitted 2020-05-28; First posted 2020-06-01 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Melatonin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Participants in this group, in addition to receiving the usual treatment of COVID-19, will receive a 9 mg dose of melatonin for seven to ten nights.
  Interventions: Drug: Melatonin; Drug: The usual treatment
- Control Group (Active Comparator): Participants in this group will receive the usual treatment of COVID-19
  Interventions: Drug: The usual treatment

INTERVENTIONS:
Drug: Melatonin — Participants in this group, in addition to receiving the usual treatment of COVID-19, will receive a 9 mg dose of melatonin for seven to ten nights.
  Arms: Test Group
Drug: The usual treatment — Participants in this group will receive the usual treatment of COVID-19

SUMMARY:
The leading cause of death in patients with COVID19 is a severe inflammatory response caused by a cytokine storm that results in acute respiratory distress syndrome and acute pulmonary insufficiency, as well as dysfunction of several vital organs. Therefore, preventing the occurrence of uncontrolled inflammation is the main goal of the ongoing clinical trials. Chloroquine and tocilizumab, which have the best results, are also prescribed to control inflammation. But it can be said that treatments are the main source of inflammation. Inflammasome NLRP3 is one of the mechanisms involved in many severe inflammatory disorders. Inflammatory activation has already been demonstrated by many viruses. Melatonin, on the other hand, is a hormone in the body that can inhibit Inflammation NLRP3 in addition to various anti-inflammatory effects, especially after severe inflammation. Older adults with lower levels of melatonin and children with maximum levels of melatonin are the risk groups and low-risk groups for the disease, respectively. In the present study, while measuring melatonin in patients with COVID19, its effectiveness as a treatment method along with the common antiviral drug regimen in patients with severe disease will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COVID-19 based on either ground glass appearance in chest CT scan or positive RT-PCR test for COVID-19
* Oxygen saturation drop below 93%
* Systolic blood pressure drop below 100 or blood pressure drop of 30 mm Hg from the patient's previous normal systolic blood pressure
* Fever
* Dry cough
* Positive PCR for COVID-19
* Laboratory indices include CRP and ESR indicating COVID-19

Exclusion Criteria:

* Patient dissatisfaction
* Existence of drug interactions
* Lack of proper conditions for receiving medication

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2020-05-12 (Actual); Primary Completion 2020-06-05 (Estimated); Study Completion 2020-09-25 (Estimated)

PRIMARY OUTCOMES:
Melatonin | up to 10 days
  Immune system modulator. The amount of it is determined by laboratory methods

SECONDARY OUTCOMES:
Inflammatory cytokines | up to 10 days
  is a type of signaling molecule (a cytokine) that is secreted from immune cells like helper T cells (Th) and macrophages, and certain other cell types that promote inflammation which is measured by serological or analyzer method
C-reactive protein (CRP) | up to 10 days
  C-reactive protein (CRP) is a protein made by the liver that measured by serological or analyzer method
Cough | up to 10 days
  A sudden, audible expulsion of air from the lungs through a partially closed glottis, preceded by inhalation. It is a protective response that serves to clear the trachea, bronchi, and/or lungs of irritants and secretions that measured by Physical examination.
Oxygen saturation of the blood | up to 10 days
  Oxygen saturation of the blood will measure by pulse oximeter
ESR | up to 10 days
  Red blood cell sedimentation rate will measure by Autoanalyzer
Radiological Treatment Response | up to 10 days
  Radiological Treatment Response (CT scan), more than 50% reduction in the affected area
Inflammatory route | up to 10 days
  Cellular pathway active in inflammation

CONTACTS AND LOCATIONS:
Locations (1):
- Mohammad Sadegh Bagheri Baghdasht, Tehran, Iran